CLINICAL TRIAL: NCT03051230
Title: Vascular Cell Activation Throughout Ovarian Hyperstimulation for In Vitro Fertilisation: Role of Cell-Derived Microparticles in the Adverse Outcomes
Brief Title: Vascular Cell Activation, Cell-Derived Microparticles and In Vitro Fertilisation, and In Vitro Fertilisation
Acronym: PREDHSO
Status: Completed | Type: Observational
Sponsor: Poissy-Saint Germain Hospital (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Principal Investigator, Antoine Torre, Medical Doctor, Poissy-Saint Germain Hospital
Other Study IDs: PREDHSO
Record Dates: First submitted 2017-02-01; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Infertility; Hyperstimulation Syndrome, Ovaian; Thrombosis
Keywords: Blood Coagulation Disorders; Cell-Derived Microparticles; Superovulation; Fertilization in Vitro; Biomarkers
MeSH Terms: conditions — Infertility; Thrombosis; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After platelet removal, serum samples will be frozen stored before being processed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Studied group: Women exposed to ovarian hyperstimulation for In Vitro fertilisation

SUMMARY:
Introduction: Ovarian hyperstimulation syndrome (OHSS) is an iatrogenic phenomenon, poorly understood and difficult to predict, complicating intense ovarian stimulation cycle. The most severe symptoms, which associate vascular permeability disorders and hypercoagulability, occur in 0.2 to 1% of the cases and often require intensive care.

Activation of endothelial, platelet, erythrocyte or leukocyte cells trigger the release of small specific vesicles, called microparticles, used as markers.

Classically leading to endothelial dysfunction and hypercoagulability, the endothelial activation phenomenon could constitute the main cause of OHSS or help predict its severity, as established for various other diseases (cerebral stroke, infarct and lupus…). However, so far, this endothelial activation role has never been studied.

Objectives:

Evaluate the serum level of microparticles as a predictor of adverse outcomes; correlate it to hypercoagulability and changes of endothelial permeability associated with this syndrome.

Methodology: Prospective Pilote Cohort study, evaluating before and throughout the ovarian stimulation cycle (6 samples/patient), the serum modulation of:

* Endothelial activation markers (endothelial-derived microparticles, E-selectin)
* Procoagulant markers (microparticles from platelet, erythrocyte or leukocyte origin, Von Willbrand factor, thrombin-antithrombin complex, prothrombin fragment 1+2)
* Endothelial disjunction marker (soluble CD 146) A group of 50 patients will be assessed Techniques: Flow cytometry for measurement of microparticles expressing non specific (Annexin V) and cell specific surface determinants (CD 31, CD 41, CD 45 or glycophorin A). Use of commercial kits for other serum markers.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years old
* With Health Insurance
* Scheduled for their first ovarian stimulation in an IVF or ICSI program in our centre
* Whose blood samples will be collected in our hospital

Exclusion Criteria:

* Suffering or having suffered from a disease likely to alter their vascular system and thus modulate their rates of microparticles:

  * auto-immune disease (systemic lupus erythematosus26, antiphospholipid syndrome)
  * cardiovascular risk factors: cardiovascular disease history, diabetes, arterial hypertension, dyslipidemia
  * Tobacco addiction.
* Presenting a blood œstradiol rate > 5000 pg/ml at ovulation triggering (criterion of stimulation cancellation) and more generally, every patient which ovulation has not been triggered.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: Infertile volunteers, aged 18 to 35 years, with neither cardiovascular disease nor Lupus erythematosus related disease, scheduled for In Vitro fertilisation, and assessed from their day 3 basal hormonal assessment, at least to the ovarian triggering of their IVF cycle were included.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-01-02 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Quantification of Microparticles subsets from endothelial origin in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of prothrombin fragment 1+2 in the circulating blood | At day 3 of an unstimulated (i.e. natural) menstrual cycle, before IVF cycle, when basal hormonal assessments is performed for fertility work-up
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from endothelial origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of prothrombin fragment 1+2 in the circulating blood | During ovarian stimulation for IVF (first cycle), at first day of FSH stimulation
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from endothelial origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of prothrombin fragment 1+2 in the circulating blood | During ovarian stimulation for IVF (first cycle), at ovarian triggering day, i.e.when ≥ 3 ovarian follicles rich 17mm
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from endothelial origin in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of prothrombin fragment 1+2 in the circulating blood | 4 days after ovarian triggering for IVF (first cycle), at the day of embryo transfer of the Day 2 embryos
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from endothelial origin in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | 9 days after ovarian triggering for IVF (first cycle), at mid-luteal phase
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from platelet origin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of Microparticles subsets from endothelial origin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from erythrocyte origin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from leukocyte origin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Microparticles subsets from platelet origin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with flow cytometry
Quantification of Tissue Factor-Dependent Procoagulant Activity (MP-TF) in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with home made device
Quantification of Plasmin Generation Capacity (MP-PGC) in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with home made device
Quantification of Fibrin monomer in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of D-dimer in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of E-selectin in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of soluble CD 146 in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of Von Willbrand factor in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of thrombin-antithrombin complex in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device
Quantification of prothrombin fragment 1+2 in the circulating blood | 16 days after ovarian triggering for IVF (first cycle), at the day of pregnancy test
  Venipuncture for blood sampling and exam with commercial device

IPD SHARING:
Plan to Share IPD: Undecided